CLINICAL TRIAL: NCT02791256
Title: An Open-label Pilot Study of Dose Escalation of PEGASYS on Virological Response in Patients With Chronic Hepatitis C Viral Infection Showing an Early Non-response to a Standard Course of PEGASYS Plus Ribavirin
Brief Title: A Study of Peginterferon Alfa-2a Plus Ribavirin in Early Non-Responder Participants With Chronic Hepatitis C (CHC) Genotype 1, 4, 5, and 6
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18232; 2005-000198-22 (EudraCT Number)
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

ARMS (1):
- Peginterferon Alfa-2a + Ribavirin (Experimental): Participants will receive 360 microgram (mcg) of Peginterferon Alfa-2a subcutaneous (SC) once a week plus ribavirin (1000 - 1200 milligram per day [mg/day] orally as a split dose in the morning and the evening based on the participant's body weight) for 32 weeks.
  Interventions: Drug: Ribavirin; Drug: peginterferon alfa-2a

INTERVENTIONS:
Drug: Ribavirin
  Other Names: Copegus, Ro 20-9963
Drug: peginterferon alfa-2a
  Other Names: Pegasys, Ro 25-8310

SUMMARY:
This multicenter, open-label, uncontrolled study will evaluate the efficacy and safety of increasing the dose of peginterferon alfa-2a (Pegasys) in participants with Genotype 1/4/5/6 CHC and an early non-response to a standard course of peginterferon alfa-2a plus ribavirin. The study will consist of screening (4 weeks), treatment (32 weeks), and follow-up (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Participants with serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Participants had to have been receiving their first treatment for chronic hepatitis C (i.e. previously naive to any therapy) consisting of peginterferon alfa-2a plus ribavirin for 16 weeks (+/- 10 days), without reaching a negative or 2-log drop of Serum Hepatitis C Virus Ribonucleic Acid (HCV-RNA) at Week 12 of therapy as compared to pretreatment value, and must still be on therapy (no wash out)
* HCV-RNA quantifiable by a test reporting in international units
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Participants with cirrhosis or transition to cirrhosis had to have an abdominal ultrasound, computerized tomography (CT) scan, or magnetic resonance imaging (MRI) scan without evidence of hepatocellular carcinoma and a serum alpha fetoprotein (AFP) less than (<)100 nanogram pe milliliter (ng/mL) within 6 months of study entry
* Negative urine or blood pregnancy test
* Participants had to be using two forms of effective contraception during treatment and during the 6 months after treatment end
* Able to participate and to comply with the study restrictions

Exclusion Criteria:

* Women with ongoing pregnancy or who are breast feeding and male partners of women who were pregnant
* Neutrophil count <1,500 cells/cubic millimeter (mm^3) or platelet count <90,000 cells/mm^3 before initiation of the ongoing treatment regimen; or neutrophil count <750 cells/mm^3 or platelet count <50,000 cells/mm^3 at screening while still on therapy with peginterferon alfa-2a plus ribavirin
* Hemoglobin (Hgb) <12 gram per deciliter (g/dL) before initiation of the ongoing treatment regimen; or Hgb <10 g/dL at screening while still on therapy with peginterferon alfa-2a plus ribavirin for at least 12 weeks
* Serum creatinine level greater than (>)1.5 times the upper limit of normal at screening
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) other than the currently failing Pegasys plus ribavirin combination therapy less than or equal to (<=) 6 months prior to the first dose of study drug
* Positive test for hepatitis A immunoglobulin M (IgM) antibody (anti-HAV IgM Ab), hepatitis B surface antigen (HBsAg), anti-hepatitis B core IgM antibody (anti-HBc IgM Ab), anti-Human Immunodeficiency Virus antibody (anti-HIV Ab)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV
* History of bleeding from esophageal varices or other conditions consistent with decompensated liver disease, severe psychiatric disease (especially depression), severe seizure disorder, thyroid disease, immunologically mediated disease, chronic pulmonary disease, cardiac disease, major organ transplantation or other evidence of severe illness, malignancy
* Evidence of drug abuse including excessive alcohol consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Virologic Response, as measured by ultrasensitive Roche HCV TaqMan Test | Week 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving Sustained Virologic Response (SVR), as measured by ultrasensitive Roche HCV TaqMan Test | Week 56
Percentage of Participants Achieving End-of-treatment Response, as measured by ultrasensitive Roche HCV TaqMan Test | Week 32
Mean Log Change From Baseline to Week 2, 4, 8, 12, 32, and 56 in Hepatitis C Virus Ribonucleic Acid (HCV-RNA) Viral Load | Baseline, Week 2, 4, 8, 12, 32, 56
Number of Participants With Adverse Events and Serious Adverse | Baseline up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (14):
- Belgium (14):
  - Antwerp
  - Bruges
  - Brussels
  - Charleroi
  - Edegem
  - Ghent
  - Gilly
  - Haine-Saint-Paul
  - Kortrijk
  - Leuven
  - Liège
  - Namur
  - Roeselare
  - Yvoir